CLINICAL TRIAL: NCT03859570
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized Trial of Pentoxifylline or Placebo in Addition to Standard of Care for Treatment of Proteinuria in Patients With Lupus Nephritis.
Brief Title: Pentoxifylline in Lupus Nephritis
Acronym: Pentoxifylline
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study not selected to receive funding
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Ohio State University (Other); The Research Foundation for the State University of New York (Unknown); Yale University (Other)
Responsible Party: Principal Investigator, Stanley Ballou, Professor of Medicine - Case Western Reserve University, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB18-00310
Record Dates: First submitted 2019-02-22; First posted 2019-03-01 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Contracted biostatistician will be responsible for drug/placebo randomization. He will be able to conduct an early, interim data analysis following initial 30% enrollment, and will permit unblinding of subject data to the Data Safety Monitor (DSM) for reasons of safety assurance, as requested.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pentoxifylline (Experimental): Pentoxifylline and standard of care therapy
  Interventions: Drug: Pentoxifylline
- Placebo (Placebo Comparator): Placebo and standard of care therapy
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline (PTX) is a methylxanthine derivative that is a nonselective inhibitor of cyclic nucleotide phosphodiesterase (PDE). This enzyme, which has at least 5 subtypes, is responsible for inactivation of the important second messengers, Cyclic adenosine monophosphate (AMP) and cyclic guanosine monophosphate (GMP)
  Other Names: Trental
  Arms: Pentoxifylline
Drug: Placebos — Placebo
  Arms: Placebo

SUMMARY:
Glomerulonephritis is an important manifestation in about 1/2 of patients with Systemic Lupus Nephritis (SLE; lupus). Despite recent national guidelines recommending use of induction therapy with high-dose corticosteroids and immunosuppressive agents, followed by prolonged maintenance therapy, up to 1/3 of these patients continue to have active nephritis and ongoing protein in the urine (proteinuria). It has long been recognized that both the level and chronicity of proteinuria in patients with lupus nephritis are associated with disease severity and with long-term prognosis, including the possibility of progression to complete kidney failure, which may occur in about 1/4 of patients. Pentoxifylline (PTX) is an oral medication introduced 45 years ago for treatment of vascular insufficiency. It has also recently been found to reduce proteinuria in patients with diabetic nephropathy. The mechanism of this unexpected and intriguing finding is not certain, but may in part involve inhibiting the production of TNF-alpha, an inflammatory cytokine known to be present in urine and kidneys of patients with lupus nephritis. Our hypothesis is that this inexpensive, generic drug, PTX, can significantly reduce proteinuria in patients with lupus nephritis.

To test this hypothesis, we plan to initiate a 6-month, double-blind, placebo-controlled randomized clinical trial of PTX or placebo in 40 patients with active lupus nephritis. This trial will include 6-8 patients from each of 5 different academic medical centers that specialize in the treatment of lupus nephritis. Our primary objective of this trial will be to measure urine protein each month to determine the extent to which PTX is able to reduce urine protein, and how rapidly this occurs.

Concurrently, we will carefully follow these patients each month to determine whether PTX administration is also associated with stabilization of renal function, or with improvement in other manifestations of lupus, such as clinical disease activity or abnormal laboratory findings. A major secondary objective will be to explore the possible mechanism(s) whereby PTX reduces proteinuria. For this purpose, we will use the monthly urine specimens to measure TNF-alpha, and levels of several other proteins (IL-1, IL-6, IL-2, MCP-1, TGF-beta, PDGF, and IFN-alpha) that have been shown to contribute to inflammation and scarring in lupus nephritis. Comparison of levels of these inflammatory proteins with level of protein in the urine should help us to determine whether one or more of these proteins is a contributor to the severity or persistence of lupus nephritis.

This information may also allow us to learn whether repeated measurements of these proteins can serve as biomarkers to assist in the ongoing management of patients with lupus nephritis. Finally, we hope to eventually measure levels of these inflammatory proteins in blood samples from the patients, to determine if PTX treatment can suppress (or enhance) such levels, and whether these changes are associated with reduced lupus disease activity, or improvement in other manifestations of lupus. Ultimately, it is our hope that the data from this clinical trial using a generic repurposed drug will permit us to conclusively confirm that PTX can significantly reduce proteinuria in patients with lupus nephritis, which would be of great benefit for the thousands of people who suffer with this most severe type of lupus.

DETAILED DESCRIPTION:
Glomerulonephritis occurs in up to one-half of patients with systemic lupus erythematosus (SLE) and is a major cause of morbidity and mortality. Guidelines published by the American College of Rheumatology in 2012 (1) suggested a multi-targeted treatment approach that has been shown to lead to clinical remission in up to one-half of patients (2,3).

However, at least one-third of patients continue to have active disease; many of these individuals may eventually develop renal failure. Therefore, there is an unmet need for more effective therapeutic approaches for lupus nephritis (LN). Although the pathogenesis of LN is almost certainly multifactorial, the presence and persistence of immune complexes are thought to play a major role in disease pathogenesis by attracting inflammatory cells of the innate immune system, such as neutrophils and monocytes, resulting in cell activation and secretion of inflammatory cytokines, including interferon alpha, TGF-beta, IL-1, IL-6, and TNF-alpha (6-7). Pentoxifylline (PTX) is a nonselective phosphodiesterase inhibitor with minimal toxicity. It has been in clinical use since 1972 for treatment of patients with intermittent claudication secondary to peripheral vascular disease. This generic drug has also recently been increasingly used off-label for several other conditions, including patients with diabetic nephropathy, in whom the unexpected finding of significant reduction of proteinuria has been repeatedly demonstrated (34-38). The mechanism of this phenomenon is unclear, although experimental studies in animals and humans have observed suppression of inflammatory cytokine production following PTX administration (24-28). In LN, 2 small, uncontrolled observational studies of PTX reported reduction in proteinuria following 2-6 months of treatment with PTX (8,9). The level and chronicity of proteinuria have long been associated with disease prognosis in patients with LN (10). Thus, a novel treatment that could significantly and persistently reduce or even eliminate proteinuria could result in substantial improvement in the long-term outcome of patients with this most serious manifestation of SLE.

ELIGIBILITY:
Inclusion criteria:

1. Patients 18 and older, who meet the 1997 update of the1982 criteria for classification of systemic lupus erythematosus and have established lupus nephritis as documented by any of the following:

   1. Kidney biopsy documenting class II, III, IV, or V (RPS/ISN 2004) lupus nephritis within 3 years or
   2. Abnormal urine protein excretion on 2 occasions, at least 2 weeks apart, characterized by more than 500 mg urine protein, quantitated either by 24-hour urine collection or by urine protein/creatinine ratio (UPCR) more than 0.5 mg/mg, measured on a first void morning specimen, in the absence of other glomerulopathies; or
   3. Abnormal urine sediment, containing more than 5 RBC, more than 5 WBC, or cellular casts on 2 occasions, at least 2 weeks apart, in the absence of infection, concurrent menstruation, anatomic genitourinary abnormalities, or pathologic disorders other than lupus nephritis.
2. Absence of changes in immunosuppressive agents or dose of immunosuppressive agents administered during the 2 months before enrollment. Patients with newly-diagnosed lupus nephritis will not be invited to participate until after they have completed 6 months of initial induction therapy.
3. Unless contraindicated, patients will be required to be taking an ACE inhibitor or ARB, with stable dose for at least 1 month prior to enrollment. Patients with intolerance of ACE/ARB therapies will be eligible to participate, but will be analyzed separately, as indicated in the trial synopsis.
4. Urine protein more than 500 mg/24 hours and/or UPCR more than 0.5 mg/mg at time of baseline.
5. Willingness to remain on stable immunosuppressive drugs for the 6-month duration of the study unless safety issues arise.
6. The SELENA-SLEDAI will be measured at screening but no minimal SLEDAI score will be required for inclusion.
7. Although kidney biopsy is not required for enrollment in this clinical trial, the standard of care at all participating institutions is to recommend renal biopsy for all patients with lupus nephritis, and generally at least 75% of such patients at each participating institution will be expected to have had this procedure. Subjects who qualify for this study according to clinical criteria noted in 1b and 1c above must be confirmed to have lupus nephritis, and no other renal disorder, by the site PI, prior to enrollment.

Exclusion criteria:

1. History of retinal, cerebral, or peptic ulcer hemorrhage within 3 months prior to enrollment
2. Current use of warfarin, long-acting heparin, or an oral anti-coagulant (other than low dose aspirin)
3. Pregnancy or currently breast-feeding
4. History of theophylline, pentoxifylline, or caffeine allergy
5. Currently taking theophylline-containing medications
6. Malignancy within 2 years, other than basal cell carcinoma
7. Congestive heart failure, class III or IV
8. Abnormal AST/ALT, more than 2 times ULN
9. Obstructive uropathy
10. Acute kidney injury defined as greater than 50% decrease in GFR within 30 days prior to screening.
11. Myocardial infarction, percutaneous coronary intervention, coronary bypass graft surgery, or unstable angina within 6 months prior to screening
12. BP greater than 150/95 on 2 measurements in the sitting position after 5 minutes of rest, using a manual BP cuff
13. Known diagnosis of diabetes mellitus or hemoglobin A1c greater than 8.0
14. Current (within 3 months) GFR less than 30 mL/min
15. Surgery within 3 months prior to enrollment
16. Concurrent diagnosis of antiphospholipid syndrome (APS), or presence of APS antibodies on 2 occasions, more than 12 weeks apart.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Level of proteinuria | 9 months
  Level of proteinuria measured as the protein/creatinine ratio on a morning first void specimen, recorded longitudinally at monthly intervals from baseline to 6 months, and from urine specimens provided monthly for 3 months following the 6 month study termination visit.

SECONDARY OUTCOMES:
Histopathologic subclass | 6 months
  The effect of Pentoxifylline on proteinuria relative to disease duration and histopathologic subclass.We will stratify these subjects in to 3 groups: class II, class III/IV, and class V. Given the relatively low expected frequency of class II (about 20%) and class V (about 10%), and the small total number of subjects, we will likely only be able to observe trends in responses of proteinuria to Pentoxifylline treatment in the 3 groups, without observing significant differences between groups.
Serum albumin | 6 months
  Longitudinal changes in serum albumin over 6 months
Glomerular Filtration Rate | 6 months
  Longitudinal changes in glomerular filtration rate (GFR)
Serologic markers | 6 months
  Longitudinal changes in serologic markers including anti-DNA, complement component 3 (C3), and complement component 4(C4)
SELENA-Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) Instrument Score | 6 months
  Longitudinal changes in SELENA-SLEDAI (Systemic Lupus Erythematosus Disease Activity Index) Instrument Score. This tool is a cumulative and weighted index used to assess disease activity across 24 different disease descriptors in patients with Systemic Lupus Erythematosus.This assessment can be completed to objectively assess the patient's current state of disease. The descriptors with a weight of 8 are seizure, psychosis, organic brain syndrome, visual disturbance, cranial nerve disorder, lupus headache, cerebrovascular accident, and vasculitis. The descriptors with a weight of 4 are arthritis, myositis, urinary casts, hematuria, proteinuria, and pyuria. The descriptors with a weight of 2 are rash, alopecia, mucosal ulcers, pleurisy, pericarditis, low complement, and increased DNA binding. The descriptors with a weight of 1 are fever, thrombocytopenia, and leukopenia.
Longitudinal changes in patient global activity score | 6 months
  This score measures the disease activity from the patient's perspective. It is measured from 0 to 10 with 10 being the worst.
Longitudinal changes in physician global activity score | 6 months
  This score measures the disease activity from the physician's perspective.It is measured from 0 to 10 with 10 being the worst.
Prednisone dose | 6 months
  Longitudinal changes in prednisone dose (and total cumulative prednisone dose)
Serum and urinary cytokine levels | 6 months
  Correlation between serum and urinary cytokine levels (Tumor necrosis factor(TNF-alpha), Interleukin 1 (IL1), Interleukin 6 (IL6), Interleukin 2 (IL-2), Monocyte chemoattractant protein -1 (MCP-1), Transforming growth factor beta(TGF-beta), Interferon alpha (IFN-alpha), and Platelet-derived growth factor (PDGF) and changes in urinary protein excretion at baseline and at 1, 2, 3, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Ballou, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- Metrohealth Medical Center, Cleveland, Ohio, United States